CLINICAL TRIAL: NCT00955513
Title: A Randomized, Double-blind, Multi-center, Placebo-controlled, 3-treatment Arm, Parallel Group Study to Evaluate the Efficacy and Safety of Diclofenac Diethylamine 2.32% Gel Applied Twice or Three Times Daily in Patients With Acute Ankle Sprain
Brief Title: Evaluate the Efficacy and Safety of Diclofenac Diethylamine 2.32% Gel Applied Twice or Three Times Daily in Patients With Acute Ankle Sprain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VOPO-P-307
Record Dates: First submitted 2009-08-07; First posted 2009-08-10 (Estimated); Results first posted 2011-01-26 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2011-01

CONDITIONS: Grade I/II Ankle Sprain
Keywords: Ankle sprain; soft tissue injury
MeSH Terms: conditions — Ankle Injuries; Soft Tissue Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- diclofenac diethylamine gel 2.32% gel twice a day (Experimental): drug
  Interventions: Drug: diclofenac diethylamine gel 2.32%
- diclofenac diethylamine gel 2.32% gel three times a day (Experimental): drug
  Interventions: Drug: diclofenac diethylamine gel 2.32%
- placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: diclofenac diethylamine gel 2.32% — diclofenac diethylamine gel 2.32% twice a day
  Arms: diclofenac diethylamine gel 2.32% gel twice a day
Drug: diclofenac diethylamine gel 2.32% — diclofenac diethylamine gel 2.32% three times a day
  Arms: diclofenac diethylamine gel 2.32% gel three times a day
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
The main purpose of this trial is to compare the efficacy and safety of diclofenac diethylamine 2.32% gel applied twice (b.i.d) or three times a day (t.i.d.) with placebo in the treatment of acute ankle sprains (distortions).

ELIGIBILITY:
Inclusion Criteria:

1. Acute sprain of the lateral ankle, Grade I-II .

Exclusion Criteria:

1. Any concurrent injury affecting the lower extremities that is painful at rest or on movement, or could affect the mobilization of the patient.
2. Topical analgesic or anti-inflammatory treatment over the previous month in the area to be treated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Gilching
  - Novartis Investigative Site, Grünwald
  - Novartis Investigative Site, München

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 6 centers in Germany. Recruitment commenced in July 2009 and completed in December 2009.
Groups:
- Diclofenac Diethylamine Gel 2.32% Gel. Applied 2 Times a Day; Diclofenac Diethylamine Gel 2.32% Gel. Applied 3 Times a Day: drug
- Placebo. Applied 3 Times a Day.: placebo
Period: Overall Study
Arm/Group | Diclofenac Diethylamine Gel 2.32% Gel. Applied 2 Times a Day | Diclofenac Diethylamine Gel 2.32% Gel. Applied 3 Times a Day | Placebo. Applied 3 Times a Day.
Started | 80 | 80 | 82
Completed | 79 | 78 | 79
Not Completed | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diclofenac Diethylamine Gel 2.32% Gel. Applied 2 Times a Day | Diclofenac Diethylamine Gel 2.32% Gel. Applied 3 Times a Day | Placebo. Applied 3 Times a Day. | Total
Number analyzed (Participants) | 80 | 80 | 82 | 242
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 80 | 77 | 81 | 238
  >=65 years | 0 | 3 | 1 | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 30.9 (11.4) | 32.2 (13.7) | 34.0 (12.9) | 32.4 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 31 | 28 | 90
  Male | 49 | 49 | 54 | 152
Region of Enrollment [Number; unit: participants]
  Germany | 80 | 80 | 82 | 242

OUTCOME MEASURES:

1. Primary Outcome: Measure: Pain on Movement on Day 5 (Change From Baseline).
Description: Visual analog scale (0 to 100 mm) A greater change from baseline equates to a better outcome.
Time Frame: baseline and day 5
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac Diethylamine Gel 2.32% Gel. Applied 2 Times a Day | Diclofenac Diethylamine Gel 2.32% Gel. Applied 3 Times a Day | Placebo. Applied 3 Times a Day.
Number analyzed (Participants) | 80 | 80 | 82
mm | 49.1 (19.3) | 49.7 (21.5) | 25.4 (14.8)

ADVERSE EVENTS:
Arm/Group | Diclofenac Diethylamine Gel 2.32% Gel. Applied 2 Times a Day | Diclofenac Diethylamine Gel 2.32% Gel. Applied 3 Times a Day | Placebo. Applied 3 Times a Day.
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80 | 0/82
Other Adverse Events (participants affected / at risk) | 0/80 | 1/80 | 1/82
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diclofenac Diethylamine Gel 2.32% Gel. Applied 2 Times a Day (N=80) | Diclofenac Diethylamine Gel 2.32% Gel. Applied 3 Times a Day (N=80) | Placebo. Applied 3 Times a Day. (N=82)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No